CLINICAL TRIAL: NCT04399343
Title: Dexmedetomidine for Prevention of Postoperative Delirium in Patients After Intracranial Operation for Brain Tumor: a Multicenter Randomized Controlled Trial
Brief Title: Dexmedetomidine for Prevention of Postoperative Delirium After Intracranial Operation for Brain Tumor
Acronym: DEPOD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY2019-091-02
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Central Nervous System Diseases
Keywords: dexmedetomidine; delirium; postoperative; intracranial operation; prevention
MeSH Terms: conditions — Central Nervous System Diseases; Delirium | interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Continuously intravenous infusion of dexmedetomidine hydrochloride at a rate of 0.1 μg/kg/hour (0.025 ml/kg/hour) started immediately after enrollment until 08:00 AM on the postoperative day one.
  Interventions: Drug: Dexmedetomidine
- Normal saline group (Placebo Comparator): Continuously intravenous infusion of normal saline at a rate of 0.025 ml/kg/hour started immediately after enrollment until 08:00 AM on the postoperative day one.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine hydrochloride (200 μg/2 ml) is diluted with normal saline to 50 ml and is continuously intravenous infused at a rate of 0.025 ml/kg/hour (dexmedetomidine 0.1 μg/kg/hour). The intravenous infusion begins immediately after enrollment until 08:00 AM on the postoperative day one.
  Other Names: Dexmedetomidine hydrochloride
  Arms: Dexmedetomidine group
Drug: Normal saline — Normal saline is also diluted with normal saline to 50 ml and is continuously intravenous infused at a rate of 0.025 ml/kg/hour, which is the same with the dexmedetomidine group. The intravenous infusion begins immediately after enrollment until 08:00 AM on the postoperative day one.
  Other Names: 0.9% Sodium Chloride
  Arms: Normal saline group

SUMMARY:
Postoperative delirium is common after major surgery, and is associated with adverse outcomes. Systematic reviews and meta-analyses of randomized controlled trials have shown that perioperative administration of dexmedetomidine may decrease the incidence of postoperative delirium in patients after either cardiac or non-cardiac surgery. However, neurosurgical patients are often excluded in clinical trials of postoperative delirium.

In this prospective, multicenter, randomized, double-blinded, and placebo-controlled trial with two parallel arms, ICU admitted adult patients after intracranial operation for brain tumor will be enrolled. Low-dose dexmedetomidine will be applied during the early postoperative phase. The investigators aim to evaluate the efficacy and safety of low-dose dexmedetomidine for prevention of postoperative delirium in this patient population. The primary hypothesis is that, compared to the placebo group, the prophylactic use of low-dose dexmedetomidine can decrease the incidence of postoperative delirium without significant adverse events in patients after intracranial operation for brain tumor.

DETAILED DESCRIPTION:
Postoperative delirium is common after major surgery, and is associated with adverse outcomes. However, patients with neurological illness are usually excluded from previous researches. Recently, limited studies have shown that the incidence of postoperative delirium in neurosurgical patients is approximately 20%, which is comparable to the results in other major surgery. Potential associations between postoperative delirium and adverse outcomes have also been found in neurosurgical patients. These results indicate that early prevention of postoperative delirium should be employed in this population.

As a highly selective α2-adrenergic receptor agonist, dexmedetomidine has been investigated as a preventive agent for postoperative delirium. Systematic reviews and meta-analyses of randomized controlled trials have shown that perioperative administration of dexmedetomidine may decrease the incidence of postoperative delirium in patients after either cardiac or non-cardiac surgery. However, neurosurgical patients are often excluded in clinical trials of postoperative delirium.

In this prospective, multicenter, randomized, double-blinded, and placebo-controlled trial with two parallel arms, ICU admitted adult patients after intracranial operation for brain tumor will be enrolled. Low-dose dexmedetomidine will be applied during the early postoperative phase. The investigators aim to evaluate the efficacy and safety of low-dose dexmedetomidine for prevention of postoperative delirium in this patient population. The primary hypothesis is that, compared to the placebo group, the prophylactic use of low-dose dexmedetomidine can decrease the incidence of postoperative delirium without significant adverse events in patients after intracranial operation for brain tumor.

ELIGIBILITY:
The inclusion criteria are adult patients after elective intracranial operation for brain tumor under general anesthesia and who are admitted to the ICU directly from the operating room or postoperative care unit.

The exclusion criteria include:

1. Admitted to the ICU after 22:00 PM;
2. Medical records documented preoperative history of mental or cognitive disorders including schizophrenia, epilepsy, Parkinsonism, or dementia;
3. Medical records documented inability to communicate in the preoperative period due to coma or language barrier;
4. History of drug abuse of psychoactive and anesthetic drugs;
5. Known preoperative severe sinus bradycardia (lower than 50 beats/min), sick sinus syndrome, second- or third-degree atrioventricular block, or left ventricular ejection fraction lower than 30%;
6. Serious hepatic dysfunction (Child-Pugh class C);
7. Severe renal dysfunction requiring renal replacement therapy before the surgery;
8. Allergies to ingredients or components of 5-[(1S)-1-(2,3-dimethylphenyl)ethyl]-1H-imidazole (dexmedetomidine hydrochloride);
9. American Society of Anesthesiologists (ASA) classification of IV to VI;
10. Moribund condition with low likelihood of survival for more than 24 hours;
11. Pregnancy or lactation women;
12. Current enrolment in another clinical trial;
13. Refuse to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium | From postoperative day 1 to day 5
  Postoperative delirium is defined as delirium within 5 postoperative days, which is diagnosed by the Confusion Assessment Method for the ICU (CAM-ICU) evaluated twice daily (8:00-10:00 AM, and 18:00-20:00 PM).

SECONDARY OUTCOMES:
The incidence of adverse events | From the start of study agent infusion to postoperative day 1
  Include bradycardia (defined as heart rate lower than 55 beats/min), hypotension (defined as systolic blood pressure lower than 90 mmHg), and hypoxemia (defined as pulse oxygen saturation lower than 90%)
The incidence of non-delirium complications | From the start of study agent infusion to postoperative day 28
  Include airway obstruction and apnea, respiratory failure, cardiac events, coma, epilepsy, cerebral hemorrhage or infarction, renal injury and infection
Length of stay in the ICU | From the start of study agent infusion to postoperative day 28
  Time of ICU discharge
Length of stay in hospital | From the start of study agent infusion to postoperative day 28
  Time of hospital discharge
The incidence of all-caused deaths after the operation | From the start of study agent infusion to postoperative day 28
  All of the deaths that occur after the study agent infusion

OTHER OUTCOMES:
The number of patients with the use of sedatives and analgesics | From the start of study agent infusion to postoperative day 1
  Include propofol, midazolam, opioids and nonsteroidal anti-inflammatory drugs
Pain intensity | From the start of study agent infusion to postoperative day 1
  Assessed by the critical-care pain observation tool (CPOT) with a total score of 0-8. Higher scores mean a worsening of pain.
Subjective sleep quality | From the start of study agent infusion to postoperative day 1
  Assessed by numerical rating scale (NRS) with a total score of 0-10. Higher scores mean a better sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Study Chair — Intensive Care Unit, Beijing Tiantan Hospital, Capital Medical University
Locations (1):
- Intensive Care Unit, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He X, Cheng KM, Zhang L, Gu H, Qu X, Xu Y, Ma P, Zhou JX. Dexmedetomidine for the prevention of postoperative delirium in patients after intracranial operation for brain tumours (DEPOD study): a study protocol and statistical plan for a multicentre randomised controlled trial. BMJ Open. 2020 Nov 23;10(11):e040939. doi: 10.1136/bmjopen-2020-040939. PMID 33234648